CLINICAL TRIAL: NCT04127890
Title: ELO Water In Diabetes Care For Enhancement Of Blood Sugar Control (EDEN Study) - A Double-Blinded Randomized Controlled Trial
Brief Title: ELO Water In Diabetes Care For Enhancement Of Blood Sugar Control
Acronym: EDEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Collaborators: ELO Water Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELOWater
Record Dates: First submitted 2019-10-13; First posted 2019-10-16 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus
Keywords: oxygen-enriched water
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): 1.5 L of ELO Water to be drunk daily for 24 weeks
  Interventions: Dietary Supplement: ELO Water
- Control Arm (Placebo Comparator): 1.5 L of placebo bottled drinking water to be drunk daily for 24 weeks
  Interventions: Dietary Supplement: Placebo drinking water

INTERVENTIONS:
Dietary Supplement: ELO Water — oxygen-enriched water
  Arms: Intervention Arm
Dietary Supplement: Placebo drinking water — bottled drinking water
  Arms: Control Arm

SUMMARY:
This double-blinded, randomised and controlled trial evaluates the efficacy of oxygen-enriched ELO drinking water as an adjuvant modality in diabetes care for enhancement of glycemic control in patients with Type 2 diabetes mellitus. Adults with type 2 diabetes will be randomized to drink 1.5 L of either ELO water or normal drinking water for 24 weeks. The primary outcome is improvement in glycaemic control.

DETAILED DESCRIPTION:
Global diabetes mellitus prevalence is rapidly increasing. In 2015, IDF reported that Singapore has 12.8% of its population diagnosed with diabetes mellitus, of which more than 90 percent are type 2 diabetes with underlying insulin resistance. With the aging population and increasing prevalence of obesity and sedentary lifestyles, the prevalence is expected to continue to rise.

In vitro studies demonstrated that hypoxia creates a state of insulin resistance through HIF (Hypoxia Inducible Factor) transcription factor expression in adipocytes. Insulin sensitivity was shown to improve in type 2 diabetes patients and overweight non diabetic patients placed in a hyperbaric oxygen chamber.Increased water intake has been associated with lower HbA1c in the general population , and also with lower post-prandial glucose in type 2 diabetic individuals.

This study aims to evaluate the effects of 1.5 L daily of ELO water, a drinking water enriched with molecular oxygen in a stable form, with a similar volume of bottled drinking water, on glycaemic control in adults with type 2 diabetes in Singapore.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes mellitus with HbA1c 8.0% to 11%, within the last 6 months

Exclusion Criteria:

1. Type 1 diabetes patients
2. Pregnant or lactating women
3. Comorbid conditions requiring fluid restriction to below 1.5 L daily
4. Terminal illness with life expectancy less than 1 year

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2018-05-28 (Actual)

PRIMARY OUTCOMES:
Improvement of glycaemic control | 12 weeks
  Reduction in HbA1c and fasting plasma glucose
Weight loss | 12 weeks
  Reduction in weight

CONTACTS AND LOCATIONS:
Overall Officials: Joan Khoo, Dr, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No